CLINICAL TRIAL: NCT05048537
Title: The Correlation Between the Detection Rate of 18F-FACBC PET/CT and the PSA Kinetics for Prostate Cancer Patients With Biochemical Recurrence.
Brief Title: 18F-FACBC PET/CT and the PSA Kinetics for PCa Patients With Biochemical Recurrence.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 202010009MIND
Record Dates: First submitted 2021-09-01; First posted 2021-09-17 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2021-11

CONDITIONS: Biochemical Relapse Fo Malignant Neoplasm of Prostate
Keywords: Prostate cancer; 18F-FACBC; Biochemical recurrence
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-FACBC PET/CT and the PSA kinetics for PCa patients with BCR. (Other)
  Interventions: Radiation: 18F-FACBC PET/CT

INTERVENTIONS:
Radiation: 18F-FACBC PET/CT — 10mCi 18F-FACBC IV injection, then whole body PET/CT after 4 mins

SUMMARY:
Prostate cancer (PCa) is the fifth-most common cancer for male with a seventh highest cancer-related death in Taiwan. Currently, the incidence and mortality rate are still increasing rapidly. The treatment decision planning is made up by clinical charts like Gleason score (GS), TNM stage and serum prostate-specific antigen (PSA) level. However, after definitive therapy for PCa with either external beam radiotherapy (EBRT) or radical prostatectomy (RP), up to half patients experience biochemical recurrence (BCR). Although not all patients with BCR proceed to develop disease progression, it is important to identify early lesion to initiate salvage treatment.

Anti-1-amino-3-[18F]fluorocyclobutane-1-carboxylic acid (18F-FACBC) positron emission tomography (PET) is a imaging marker for L-amino acid transport evaluation. Many cancers including PCa have up-regulated amino acid transport tied to their proliferative potential. Recently, 18F-FACBC was included in the National Comprehensive Cancer Network (NCCN) guidelines for the management of recurrent PCa patients. As we know, PSA level and PSA kinetics are valuable for the prediction of recurrence. The objective of this study is to investigate the correlation between the detection rate of 18F-FACBC PET/CT and the PSA kinetics for PCa patients with BCR.

ELIGIBILITY:
Inclusion criteria:

* PCa patients with BCR
* Serum PSA data and pathologic report
* Agreement consent

Exclusion criteria:

* Claustrophobia and unstable vital signs
* Disagreement

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — prostate cancer patients with biochemical recurrence
Enrollment: 20 (Estimated)
Dates: Start 2021-03-26 (Actual); Primary Completion 2023-11-12 (Estimated); Study Completion 2023-11-12 (Estimated)

PRIMARY OUTCOMES:
The detection rate of 18F-FACBC PET/CT | 30 minutes
  The correlation between the positive/negative results of 18F-FACBC scans and the PSA kinetics in prostate cancer patients with biochemical recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Hsien Chou, MD, Study Director — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan